CLINICAL TRIAL: NCT00136175
Title: Phase II Trial of Paclitaxel, Carboplatin and Gemcitabine in Patients With Locally Advanced Transitional Cell Carcinoma of the Bladder
Brief Title: Paclitaxel, Carboplatin and Gemcitabine in the Treatment of Patients With Advanced Transitional Cell Cancer of the Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9910
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Bladder Cancer
Keywords: Neoadjuvant chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Paclitaxel; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients with clinical stage T2 with hydronephrosis or T3 bladder cancer will receive 3 cycles of chemotherapy (200mg/m^2 paclitaxel on day 1, carboplatin on day 1, and 800 mg/m^2 gemcitabine on days 1 and 8 of each 21 day cycle).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine
- Arm II (Experimental): Patients with T4 or lymph node positive disease will receive up to 6 cycles of paclitaxel, carboplatin, and gemcitabine.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin
Drug: Gemcitabine

SUMMARY:
This trial will evaluate the efficacy and safety of combination chemotherapy (paclitaxel, carboplatin, and gemcitabine) prior to surgery in the treatment of patients with locally advanced transitional cell cancer of the bladder.

DETAILED DESCRIPTION:
This is a Phase II trial of neoadjuvant chemotherapy with paclitaxel, carboplatin and gemcitabine in the treatment of locally advanced transitional cell carcinoma of the bladder. Patients will be stratified based on extent of disease. Patients with T3, N0 disease will receive 3 cycles of chemotherapy and then proceed to cystectomy. Patients with T4 disease or any patient with N1-3 disease will receive 3 cycles of therapy followed by assessment of response. Patients with evidence of response will then receive an additional three cycles of therapy with reassessment of resectability after cycles #6. Correlative Studies: Tumor specimens obtained at initial biopsy will be assayed for expression of p53, Rb and p21.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven locally advanced (T3-4, N0 or Tany, N1-3) urothelial carcinoma of the bladder. Patients with local disease and unilateral or bilateral hydronephrosis will be eligible and included in the T3 arm of the study.
* Tumor specimens must be available for assay of molecular markers.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 2 (a measure of general well being where 0 is asymptomatic and 5 is death)
* Life expectancy of 12 weeks or more
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Patients may not have had prior systemic or intra-arterial chemotherapy and no prior radiotherapy (Patients may have received intravesicular chemotherapy).
* Evidence of distant metastasis
* Unresolved bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 1999-11; Primary Completion 2005-12 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients in Arm I with Complete Pathologic Response | 3 Cycles (63 days) of Treatment
  To assess the overall response measured as complete pathologic response and conversion to resectability of the combination of paclitaxel, carboplatin and gemcitabine in patients with locally advanced transitional cell carcinoma of the bladder.
Percentage of Patients in Arm II that Obtain to Resectable Disease | 6 Cycles (126 days) of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States